CLINICAL TRIAL: NCT02503059
Title: Etanercept Survival in Elderly Population
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPA-ETA-2014-01
Record Dates: First submitted 2015-07-08; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the 3-year survival of etanercept in patients over 60 years with psoriasis in moderate / severe plaque and the reasons that led to the abandonment. Besides factors that might have had a positive or negative influence on adherence to treatment and analysis of efficacy (PASI 75) and safety will be identified.

All variables were collected through retrospective review of medical records of patients dermatology unit are made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate / severe psoriasis (with / without psoriatic arthritis,PAs) defined by: PASI(Psoriasis Area and Severity Index)> 10 and / or BSA(Body Surface Area)> 10% and / or DLQI(Dermatology Life Quality Index)> 10
* PASI> 10 and / or BSA(Body Surface Area)> 10% and / or DLQI(Dermatology Life Quality Index)> 10
* Over 60 years of age at the start of treatment
* Receiving etanercept at any time
* Available history in the Dermatology

Exclusion Criteria:

* Patients with insufficient clinical data in the medical record

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 60 who received etanercept for the treatment of moderate / severe psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
primary ineffectiveness in patients with etanercept treatment | 24 weeks
  Number of participants not achieve PASI 50 response at 12 weeks
Secondary ineffectiveness in patients with etanercept treatment | 24 weeks (duration of treatment with etanercept)
  Number of participants with Poor adherence to treatment with etanercept",
Ineffectiveness of treatment in localized lesions in patients with etanercept treatment | 24 weeks(duration of treatment with etanercept)
  Despite having achieved a good response PASI no improvement in critical injuries
primary ineffectiveness in patients with etanercept treatment | 24 weeks
  Number of participants not achieve PASI 75 response at 24 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events during treatment with etanercept | 24 weeks
Number of participants with disease remission | 24 weeks
number of participants with Poor adherence to treatment with etanercept | 24 weeks
number of participants with Conditions requiring hospitalization and / or surgery | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Herrera Ceballos, MD, Study Director — H.U. Virgen de la Victoria
Locations (5):
- Spain (5):
  - Hospital Clinic, Barcelona, Barcelona
  - H.U. Reina Sofía, Córdoba, Córdoba
  - Hospital de Andújar, Jaén, Jaén
  - Hospital la Paz, Madrid, Madrid
  - H.U. Virgen de la Victoria, Málaga, Málaga